CLINICAL TRIAL: NCT06790472
Title: Assessing the Glycemic Impact of an Online Lifestyle Intervention Using CGM (Continuous Glucose Monitoring). a Pilot Study.
Brief Title: Metabolic Wellness and CGM
Status: Enrolling by invitation | Type: Observational
Sponsor: David Kerr (Other)
Collaborators: William Marsh Rice University (Other); Abbott Diabetes Care (Industry)
Responsible Party: Sponsor-Investigator, David Kerr, Senior Investigator, Diabetes and Digital Health Equity, Palo Alto Medical Foundation
Organization: Palo Alto Medical Foundation (Other)
Other Study IDs: 2024.055-1
Record Dates: First submitted 2024-09-25; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-09

CONDITIONS: Cardiometabolic Risk Factors
Keywords: Lifestyle; Online; Metabolic wellness; Cardiometabolic risk; Digital health; Continuous glucose monitoring
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SH MWP Participants (Fall 2024): Research participants will be Sutter Health employees and their dependents who enroll in the MWP and are invited to participate in a research study about the program. Over 8 weeks, program participants will engage in an online program focusing on evidence-based lifestyle interventions which include education related to food choices, physical activity, sleep, and stress guidance.
  Interventions: Behavioral: Online Lifestyle Intervention; Device: Continuous Glucose Monitoring

INTERVENTIONS:
Behavioral: Online Lifestyle Intervention — The Metabolic Wellness Program (MWP) is an established 8-week program that provides participants with health education videos and webinars that focus on evidence-based nutrition, fitness, sleep, and stress intervention, including with CGM, allowing participants to monitor their real-time glucose data and to learn which lifestyle choices are best for their glycemic control and personal metabolic health. The program is also intended to help healthy participants maintain their metabolic health and lower their potential risk of developing cardiometabolic disease, as well as at-risk and pre-diabetic participants preventing the progression to T2D and people with established T2D reverse their condition.
Device: Continuous Glucose Monitoring — CGM measurements begin at enrollment with training provided digitally Participants will be asked to "live life as usual" whilst wearing the device with initial 10-14 day readings providing baseline data. Participants will participate in the online lifestyle program, which the investigators refer to as the "intervention stage." Participants will also receive questionnaires on behavior change at the beginning of week 5. During the final two weeks of the program (weeks 7-8), the final 10-14 days of CGM will be used as comparison data with baseline information.

SUMMARY:
The primary objective of this study is to determine the impact of participating in an online lifestyle intervention program on glycemic control as measured by Continuous Glucose Monitoring (CGM), with the primary outcome being the time-in-range (TIR) between 70 and 140 mg/dl comparing before the intervention, at the start of the program (week 1), and after the intervention (week 8).

DETAILED DESCRIPTION:
The Metabolic Wellness Program (MWP) is an established 8-week program that provides participants with digitally delivered health education focusing on metabolic health. The program content is based on nutrition education, promotion of physical activity, stress reduction and the need for quality sleep. The MWP also includes the use of continuous glucose monitoring (CGM), The MWP is aimed at adults with pre-existing type 2 diabetes (T2D), prediabetes and also individuals who wish to retain their metabolic health. (More information about the program is available here: https://www.sutterhealth.org/classes-events/the-metabolic-wellness-program-34466

To evaluate the success (or otherwise) of the MWP, the aim of this pilot study is to assess the impact of participating in the MWP on glycemic control, with the primary outcome being the time-in-range between 70 and 140 mg/dl measured by CGM. Data from this pilot study will provide evidence for a larger future randomized controlled trial (RCTs).

The secondary objectives are to:

* Examine additional changes in CGM variables comparing before (at baseline)and after the intervention (at week 8 and at 3 months post-intervention) Examine changes in self-reported behavior changes related to food choices, physical activity, sleep quality, and stress levels.
* Examine changes in lab values (if available as part of routine clinical care from the previous 12 months and up to 6 months after the program): and
* Examine engagement with the program, engagement with CGM, and satisfaction with the program

ELIGIBILITY:
Inclusion Criteria:

* Adults who are enrolled in the MWP
* Adults ≥ 18 years of age at enrollment.
* Willing to wear a CGM device.
* Sutter Health employee or employee's dependent enrolled in SutterSelect Employee Medical Benefits

Exclusion Criteria:

* Pregnancy
* Taking insulin
* Chronic kidney disease and on dialysis
* Any active clinically significant disease or disorder which, in the investigator's opinion, could interfere with participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be adults who respond to email, newsletters and MHO messaging advertisements addressed to Sutter Health workforce members.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-11 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control (Time-in-Range) | Baseline and Weeks 2, 7-8
  Time-in-range (TIR) between 70 and 140 mg/dl as measured by CGM.

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto Medical Foundation, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not have approval to share IPD for this project.

REFERENCES:
- See also: Sutter Health Metabolic Wellness Program — https://www.sutterhealth.org/services/primary/metabolic-wellness-program